CLINICAL TRIAL: NCT06308978
Title: A Phase 1 Study of FT819 in B-cell Mediated Autoimmune Disease
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Fate Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: FT819-102
Record Dates: First submitted 2024-03-06; First posted 2024-03-13 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Antineutrophilic Cytoplasmic Antibody (ANCA)- Associated Vasculitis (AAV); Idiopathic Inflammatory Myositis (IIM); Systemic Sclerosis (SSc); Systemic Lupus Erythematosus (SLE)
Keywords: FT819; Fate Therapeutics; Idiopathic inflammatory myositis (IIM); Systemic lupus erythematosus (SLE); Systemic sclerosis (SSc); Antineutrophilic cytoplasmic antibody (ANCA)-associated vasculitis (AAV); Allogeneic CAR-T; CD19-Targeted Therapy; Cell Therapy for Autoimmune Diseases; B-Cell Depletion in Autoimmune Disease; Phase 1 Clinical Trial; Allogeneic CAR cells; Autoimmune Diseases; A Phase 1 Study of FT819 in B-cell Mediated Autoimmune Diseases
MeSH Terms: conditions — Anti-Neutrophil Cytoplasmic Antibody-Associated Vasculitis; Myositis; Scleroderma, Systemic; Lupus Erythematosus, Systemic; Autoimmune Diseases | interventions — fludarabine; fludarabine phosphate; Cyclophosphamide; Bendamustine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Regimen A (Single dose with AMP) (Experimental)
  Interventions: Drug: FT819; Drug: Fludarabine; Drug: Cyclophosphamide; Drug: Bendamustine
- Regimen B (Single-dose without AMP, with background therapy) (Experimental)
  Interventions: Drug: FT819
- Regimen C (Two-dose with AMP) (Experimental)
  Interventions: Drug: FT819; Drug: Fludarabine; Drug: Cyclophosphamide; Drug: Bendamustine
- Regimen D (Two-dose without AMP, with background therapy) (Experimental)
  Interventions: Drug: FT819
- Regimen B1 (Single-dose without AMP, background therapy temporarily suspended) (Experimental)
  Interventions: Drug: FT819

INTERVENTIONS:
Drug: FT819 — FT819 will be administered as intravenous (IV) infusion at planned dose levels.
Drug: Fludarabine — Fludarabine will be administered as an IV infusion at planned dose levels.
  Other Names: FLUDARA
  Arms: Regimen A (Single dose with AMP); Regimen C (Two-dose with AMP)
Drug: Cyclophosphamide — Cyclophosphamide will be administered as an IV infusion at planned dose levels.
  Other Names: CYTOXAN
  Arms: Regimen A (Single dose with AMP); Regimen C (Two-dose with AMP)
Drug: Bendamustine — Bendamustine will be administered as an IV infusion at planned dose levels.
  Arms: Regimen A (Single dose with AMP); Regimen C (Two-dose with AMP)

SUMMARY:
This is a phase 1 study designed to evaluate the safety, pharmacokinetics (PK), and anti-B-cell activity of FT819 following treatment with or without auxiliary medicinal product (AMP) in participants with moderate to severe active systemic lupus erythematosus (SLE), antineutrophilic cytoplasmic antibody (ANCA)-associated vasculitis (AAV), idiopathic inflammatory myositis (IIM), and systemic sclerosis (SSc). The study will consist of a dose-escalation stage, followed by an expansion stage to further evaluate the safety and activity of FT819.

ELIGIBILITY:
Key Inclusion Criteria:

* Age: 12 to 70 years old.
* Diagnosis: Must have active B-cell mediated autoimmune disease (SLE, AAV, IIM, or SSc) confirmed by standard criteria.
* Disease Severity: Moderate to severe, requiring at least two prior treatments that were ineffective.
* Health Status: Adequate organ function to tolerate treatment.
* Consent: Able to provide informed consent or assent/obtain parental consent and comply with study procedures.

Key Exclusion Criteria:

* Pregnancy/Breastfeeding: Women must not be pregnant or nursing.
* Severe Organ Dysfunction: Significant heart, lung, liver, or kidney impairment.
* Active Infections: No recent or ongoing serious infections.
* Recent Cancer or Prior Cell Therapy: No active/recent malignancies, prior CAR T-cell therapy, or organ transplant.
* Allergies: No known allergies to study treatments.
* Weight Restriction: Must weigh at least 50 kg (110 lbs).

Ages: 12 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 244 (Estimated)
Dates: Start 2024-03-28 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2042-09-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-emergent adverse events (TEAEs) | Up to approximately 2 years
  The number of participants with TEAEs will be reported.
Number of participants with serious TEAEs | Up to approximately 2 years
  The number of participants with serious TEAEs will be reported.
Number of participants with dose-limiting toxicities (DLTs) | Up to approximately 29 days
  The number of participants with DLTs will be reported.
Recommend Phase 2 dose (RP2D) of FT819 | Up to approximately 2 years
  The RP2D will be determined.

SECONDARY OUTCOMES:
Plasma concentration of FT819 | At designated time points up to approximately 29 days
  The plasma concentration of FT819 will be determined.
Impact of treatment on quality of life | Up to approximately 2 years
  Assess changes in patient-reported health outcomes using the SF-36 survey.
Disease Activity | Up to approximately 2 years
  Evaluate improvements in disease-specific measures, such as:
  * SLE: Reduction in SLEDAI-2K score, rates of achieving DORIS, LLDAS
  * AAV: Proportion of patients achieving remission (BVAS v3) and relapse-free survival.
  * IIM: Proportion of patients achieving Myositis Response Criteria Total Improvement Score (MRC TIS major, moderate, minimal).
  * SSc: Changes in modified Rodnan Skin Score (mRSS) and lung function tests (FVC, DLCO).

CONTACTS AND LOCATIONS:
Locations (16):
- United States (11):
  - Providence Medical Foundation, Fullerton, California
  - University of California Irvine, Irvine, California
  - Children's Hospital Los Angeles Division Of Rheumatology, Los Angeles, California
  - University of California San Francisco, San Francisco, California
  - University of Minnesota Medical School, Minneapolis, Minnesota
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Montefiore Medical Center, New York, New York
  - Duke University Health System, Durham, North Carolina
  - MetroHealth, Cleveland, Ohio
  - University of Oklahoma, Oklahoma City, Oklahoma
  - Regional One Health, Memphis, Tennessee
- Hôpital La Pitié Salpêtrière, Paris, France
- Uppsala University, Uppsala, Uppland, Sweden
- United Kingdom (3):
  - Manchester University NHS Foundation Trust, Manchester, Greater Manchester
  - Cambridge University Hospitals NHS Foundation Trust, Cambridge
  - University College of London Hospitals NHS Trust (UCLH), London

IPD SHARING:
Plan to Share IPD: Undecided